CLINICAL TRIAL: NCT05869773
Title: An Open-Label, Multicenter Switch Study Evaluating Changes in Blood Pressure in Participants With Narcolepsy Switching From High-Sodium Oxybate to XYWAV
Brief Title: A Switch Study From High-Sodium Oxybate to XYWAV to Evaluate Changes in Blood Pressure in Participants With Narcolepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP258-406
Record Dates: First submitted 2023-05-12; First posted 2023-05-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Narcolepsy
Keywords: Narcolepsy Type 1; Narcolepsy Type 2; XYWAV; JZP258; Oxybate
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JZP258 (Experimental): Participants will receive 6 to 9 grams per night of JZP258 (XYWAV) for 6 consecutive weeks.
  Interventions: Drug: JZP258

INTERVENTIONS:
Drug: JZP258 — 0.5 g/ml calcium, magnesium, potassium, and sodium oxybates oral solution
  Other Names: XYWAV

SUMMARY:
The aim of this study is to quantify the change in blood pressure when participants with narcolepsy treated with high-sodium oxybate are transitioned to XYWAV, a low-sodium oxybate. The results of this study may provide health care providers (HCPs), patients, and payers with important new information regarding BP changes related to differences in sodium content between available oxybates for the treatment of narcolepsy.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be 18 to 70 years of age inclusive, at the time of signing the informed consent.
* Participants have a documented diagnosis of Type 1 or Type 2 narcolepsy that meets International Classification of Sleep Disorders (ICSD)-3 or Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria.
* Participants must have been receiving a total dose of high-sodium oxybate (eg, XYREM) of 6 to 9 g/night (inclusive) with twice-nightly dosing for a minimum of 6 consecutive weeks prior to screening.
* If currently treated with stimulants and/or alerting agents or other medications known to affect BP, participant must have been taking the same dosing regimen for at least 2 months prior to screening and agree to take the same dose throughout the study.
* If currently taking stable doses of antihypertensive therapies, participant must maintain these treatments at the same dose throughout the study unless otherwise advised by their medical care
* Participant is male or female. A female participant is eligible to participate if she is not pregnant or breastfeeding, if she is a woman of nonchildbearing potential or is a woman of childbearing potential and using a contraceptive method that is highly effective.

Key Exclusion Criteria:

* History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the participant or interfere with study assessments or the ability of the participant to complete the study based on the judgment of the investigator.
* Presence of significant cardiovascular disease or cardiovascular condition that in the investigator's opinion may jeopardize participant safety in the study, including screening ECG results.
* Presence of atrial fibrillation detected on screening electrocardiogram (ECG).
* Presence of resistant hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to End of Treatment (EOT) Visit on the 24-hour average Systolic Blood Pressure (SBP) in mmHg | Baseline, Up to 6 weeks

SECONDARY OUTCOMES:
Change from baseline to EOT Visit on the daytime average SBP in mmHg | Baseline, Up to 6 weeks
Change from baseline to EOT Visit on the seated resting average SBP in mmHg | Baseline, Up to 6 weeks
Change from baseline to EOT Visit on the nighttime average SBP in mmHg | Baseline, Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (43):
- United States (31):
  - Science 37, Culver City, California
  - M3 Wake Research, Encino, California
  - So Cal Clinical Research, Huntington Beach, California
  - Long Beach Research Institute, Lakewood, California
  - Stanford School of Medicine, Redwood City, California
  - TriValley Sleep Center, San Ramon, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - FWD Clinical Research, Boca Raton, Florida
  - Meris Clinical Research, LLC, Brandon, Florida
  - Ocean Wellness Center, Miami, Florida
  - Serenity Research Center LLC, Miami, Florida
  - Florida Pediatric Research Institute, LLC, Orlando, Florida
  - Sleep Practitioners, LLC, Macon, Georgia
  - Saltzer Medical Group, Nampa, Idaho
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Neurocare, Inc, Newton, Massachusetts
  - Sparrow Health System, Lansing, Michigan
  - Bryan Medical Center, Lincoln, Nebraska
  - Henderson Clinical Trials LLC, Henderson, Nevada
  - Advanced Respiratory and Sleep Medicine, PLLC, Huntersville, North Carolina
  - Intrepid Research, LLC, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience, Dublin, Ohio
  - OHSU Hospital, Portland, Oregon
  - Abington Neurological Associates, LTD, Abington, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Velocity Clinical Research, Greenville, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem
  - Private Practice RESPISOM Namur, Namur
- France (3):
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble, Isere
  - CHU Nantes - Hôtel Dieu, Nantes, Loire Atlantique
- Italy (3):
  - IRCCS Istituto de Scienze Neurologiche di Bologna (ISNB), Bologna
  - Ospedale San Raffaele (San Raffaele Turro), Milan
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
- Spain (4):
  - Hospital Universitario Araba - Sede Santiago, Vitoria-Gasteiz, Alava
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General de Castellon, Castellon
  - Hospital Universitario Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White WB, Kovacs RJ, Alexander JK, Baranak C, Nichols DA, Fuller DS, Dai J, Whalen M, Ajayi A, Hutchinson B, Dauvilliers Y, Somers VK. Effects of High- Versus Low-Sodium Oxybate on Blood Pressure in Patients With Narcolepsy. Hypertension. 2025 Dec;82(12):2162-2171. doi: 10.1161/HYPERTENSIONAHA.125.25730. Epub 2025 Oct 15. PMID 41090230